CLINICAL TRIAL: NCT05306223
Title: A Pragmatic Randomized Controlled Trial to Evaluate the Efficacy and Safety of an Oral Short-course Regimen Including Bedaquiline for the Treatment of Patients With Multidrug-resistant Tuberculosis in China
Brief Title: A Study of an Oral Short-course Regimen Including Bedaquiline for the Treatment of Participants With Multidrug-resistant Tuberculosis in China
Acronym: PROSPECT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Chest Hospital (Other)
Responsible Party: Principal Investigator, Gao Mengqiu, Director of Department of Tuberculosis, Beijing Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMC207TBC4006; TMC207TBC4006 (Other: Janssen Research & Development LLC)
Record Dates: First submitted 2022-03-23; First posted 2022-04-01 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Tuberculosis, Multidrug-Resistant
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant | interventions — bedaquiline; Levofloxacin; Linezolid; Cycloserine; Clofazimine; Pyrazinamide; Prothionamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bedaquiline-containing Short-course Regimen (SCR) (Experimental): Participants will receive an oral dose of bedaquiline 400 milligrams (mg) once daily for first 2 weeks followed by bedaquiline 200 mg thrice a week for 22 weeks (with at least 48 hours between doses) in combination with oral doses of levofloxacin (LFX) up to 1000 mg (weight-based), cycloserine (CS) up to 750 mg (weight-based), clofazimine (CFZ) 100 mg daily for 40 weeks and linezolid [LZD] 600 mg daily for at least 24 weeks . If a participant is still sputum culture-positive for Mycobacterium tuberculosis by Week 16, bedaquiline treatment will be extended from Week 24 to Week 40.
  Interventions: Drug: Bedaquiline; Drug: Levofloxacin; Drug: Linezolid; Drug: Cycloserine; Drug: Clofazimine
- Non-bedaquiline-containing Short-course Regimen (SCR) (Experimental): Participants will receive oral doses of LFX up to 1000 mg (weight-based), CS up to 750 mg (weight-based), CFZ 100 mg, Pyrazinamide (PZA) up to 2000 mg (weight-based), Protionamide (PTO) up to 800 mg (weight-based) daily for first 16 weeks and LZD 600 mg daily for at least 24 weeks.
  Interventions: Drug: Levofloxacin; Drug: Linezolid; Drug: Cycloserine; Drug: Clofazimine; Drug: Pyrazinamide; Drug: Protionamide

INTERVENTIONS:
Drug: Bedaquiline — Bedaquiline uncoated tablets will be administered orally.
  Other Names: SIRTURO
  Arms: Bedaquiline-containing Short-course Regimen (SCR)
Drug: Levofloxacin — Levofloxacin filmcoated will be administered orally
Drug: Linezolid — Linezolid tablets will be administered orally
Drug: Cycloserine — Cycloserine capsules will be administered orally.
Drug: Clofazimine — Clofazimine capsules will be administered orally.
Drug: Pyrazinamide — Pyrazinamide tablets will be administered orally.
  Arms: Non-bedaquiline-containing Short-course Regimen (SCR)
Drug: Protionamide — Protionamide enteric-coated tablets will be administered orally.
  Arms: Non-bedaquiline-containing Short-course Regimen (SCR)

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of an oral bedaquiline-containing multidrug-resistant tuberculosis (MDR-TB) short-course regimen (SCR) compared to an oral SCR not including bedaquiline at the end of treatment in participants with pulmonary MDR-TB in China.

ELIGIBILITY:
Inclusion Criteria:

* Has a positive sputum Mycobacterium tuberculosis culture from a test performed at screening
* Has microbiological confirmation of rifampicin resistance by GeneXpert and to isoniazid (INH) via molecular drug-susceptibility testing (DST) showing katG mutation
* Has a chest imaging result compatible with a diagnosis of pulmonary Tuberculosis (TB)
* Agrees to use effective contraception during the 40-week study treatment phase. A female participant must be: of nonchildbearing potential; of childbearing potential and practicing effective methods of contraception during the 40-week study treatment phase
* Is willing to undergo human immunodeficiency virus (HIV) testing

Exclusion Criteria:

* Has received prior treatment with bedaquiline
* Has prior exposure to at least 1 second-line drug in the regimen for at least 4 weeks
* Has any grade 3 or 4 laboratory abnormality as confirmed by a clinical expert
* Has a known allergy or intolerance to bedaquiline or other drugs in the regimen
* Is infected with a strain of nontuberculous mycobacteria
* Is HIV-positive

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2025-08-08 (Estimated); Study Completion 2025-08-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with a Favorable Treatment Outcome at the End of Treatment | At the end of treatment (Week 40)
  Percentage of participants with a favorable treatment outcome at the end of treatment will be reported. A participant's outcome will be classified as favorable if their last 3 culture results by the end of treatment are negative unless they have previously been classified as unfavorable. These 3 cultures must be taken on separate visits; the latest of which being no more than 8 weeks prior to the end of treatment.

SECONDARY OUTCOMES:
Percentage of Participants with a Favorable Treatment Outcome at 48 Weeks Post the End of Treatment | At 48 weeks post the end of treatment (Week 88)
  Percentage of participants with a favorable treatment outcome at 48 weeks post the end of treatment will be reported. A participant's outcome will be classified as favorable if their last 3 culture results by the end of treatment are negative unless they have previously been classified as unfavorable. These 3 cultures must be taken on separate visits; the latest of which being no more than 8 weeks prior to the end of treatment.
Percentage of Participants Achieving Treatment Success at the end of Treatment | At the end of treatment (Week 40)
  Percentage of participants achieving treatment success at the end of treatment will be reported. Treatment success is achieved if participants completed their prescribed tuberculosis (TB) treatment; or if their last 3 culture results are negative by the end of treatment, these 3 cultures must be taken on separate visits and should be after the initial 6-month treatment period.
Percentage of Participants with a Modified Favorable Treatment Outcome at the end of Treatment and at 48 Weeks Post end of Treatment | At the end of treatment (Week 40) and at 48 weeks post end of treatment (Week 88)
  Percentage of participants with a modified favorable treatment outcome at the end of treatment and at 48 weeks post end of treatment will be reported. A participant's treatment outcome will be classified as modified favorable if their last 2 culture results by the end of treatment are negative unless they have previously been classified as unfavorable. These 2 cultures must be taken on separate visits; the latest of which being no more than 8 weeks prior to the end of treatment.
Percentage of Participants Experiencing All-cause Mortality | Up to Week 88
  Percentage of participants experiencing all-cause mortality will be reported.
Percentage of Participants Experiencing Grade 3 or Greater Treatment-emergent Adverse Events (TEAEs) During Study Treatment and Follow-up | During study treatment and follow-up (From Week 1 up to Week 88)
  Percentage of participants experiencing grade 3 or greater TEAEs during study treatment and follow-up will be reported. An adverse event (AE) is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. TEAEs are defined as any event that begins or worsens in severity after initiation of study drug through to the end of study. An assessment of severity grade will be made using the following 5 general categorical descriptors based on division of acquired immunodeficiency syndrome (AIDS) grading for AE severity assessment. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening, and Grade 5= Death.
Percentage of Participants Experiencing TEAEs | From Week 1 up to Week 88
  Percentage of participants experiencing TEAEs will be reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. TEAEs are defined as any event that begins or worsens in severity after initiation of study drug through to the end of study.
Percentage of Participants with TB Relapses and Re-infections During the Treatment-free Follow-up Phase | During the treatment-free follow-up phase (Up to 48 weeks)
  Percentage of participants with TB relapses and re-infections during the treatment-free follow-up phase will be reported.
Percentage of Participants Whose Isolates Develop Resistance to Bedaquiline and Other Drugs Used in the Regimen | Up to Week 88
  Percentage of participants whose isolates develop resistance to bedaquiline and other drugs used in the regimen will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Mengqiu Gao, Principal Investigator — Beijing Chest Hospital
Locations (17):
- China (17):
  - Beijing Chest Hospital, Beijing
  - The Eighth Medical Center of PLA General Hospital, Beijing
  - Changsha Central Hospital, Changsha
  - Public health clinical medical center of Chengdu, Chengdu
  - Chongqing Public Health Medical Center, Chongqing
  - The Pulmonary Hospital of Fuzhou in Fujian Province（The tuberculosis control and prevention Hospital of Fuzhou in Fujian Province）, Fuzhou
  - Guiyang Public Health Clinical Center, Guiyang
  - Anhui Chest Hospital, Hefei
  - Infectious Disease Hospital of Heilongjiang Province, Heilongjiang
  - Jiamusi Tumor Hospital, Jiamusi
  - Jiangxi Chest Hospital, Jiangxi
  - Shandong public health clinical center, Shandong
  - Shanghai Pulmonary Hospital, Shanghai
  - Shenyang Chest Hospital, Shenyang
  - Wuhan Pulmonary Hospital, Wuhan
  - Xi'an Chest Hospital, Xi'an
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang

REFERENCES:
- [Derived] Gao J, Gao M, Du J, Pang Y, Mao G, Lounis N, Bakare N, Jiang Y, Zhan Y, Liu Y, Li L; Trial Team. A pragmatic randomized controlled trial to evaluate the efficacy and safety of an oral short-course regimen including bedaquiline for the treatment of patients with multidrug-resistant tuberculosis in China: study protocol for PROSPECT. Trials. 2024 Apr 1;25(1):227. doi: 10.1186/s13063-024-07946-9. PMID 38561815